CLINICAL TRIAL: NCT01714544
Title: An Open-Label, Multicenter Study of the Efficacy of Cloderm® Cream (Clocortolone Pivalate, 0.1%) in the Treatment of Moderate Plaque Psoriasis for 28 Days
Brief Title: Study of the Efficacy of Cloderm® Cream in the Treatment of Moderate Plaque Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Promius Pharma, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDC1201
Record Dates: First submitted 2012-10-23; First posted 2012-10-26 (Estimated); Results first posted 2014-07-23 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-06

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cloderm Cream (Experimental): Cloderm (clocortolone pivalate) Cream 0.1%, twice daily for 28 days
  Interventions: Drug: Cloderm Cream

INTERVENTIONS:
Drug: Cloderm Cream

SUMMARY:
The purpose of this study is to determine whether Cloderm Cream is effective for topical treatment of moderate psoriasis over 28 days.

DETAILED DESCRIPTION:
The objective of this study is to estimate the efficacy of Cloderm Cream for topical treatment of moderate plaque psoriasis over 28 days using current standards for evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Subject understands the study procedures and agrees to participate by giving written informed consent.
2. Subjects must be at least 18 years of age.
3. Subjects must present with a clinical diagnosis of stable (at least 3 months) plaque-type psoriasis.
4. Subjects with psoriasis involving 2 to 20% BSA, not including the face, scalp and intertriginous areas.
5. Subjects must have an IGA Grade of 3 at the Baseline Visit.
6. Female subjects of childbearing potential must have a negative urine pregnancy test result at Baseline (Visit 2) (test will have a sensitivity of at least 25mIU/ml for human chorionic gonadotropin) and practice a reliable method of contraception or remain sexually inactive throughout the study.

   All women of childbearing potential must be willing to undergo a urine pregnancy test at Visit 2 (Day 0), at Visit 4 (Day 14), and at Visit 5 (Day 28).
7. Subjects must be in good general health as determined by the investigator and supported by the medical history and normal or not clinically significant abnormal vital signs (blood pressure and pulse).

Exclusion Criteria:

1. Current diagnosis of unstable forms of psoriasis including guttate, erythrodermic, exfoliative or pustular psoriasis.
2. Other inflammatory skin disease that may confound the evaluation of the plaque psoriasis (e.g., atopic dermatitis, contact dermatitis, tinea corporis).
3. Presence of pigmentation, extensive scarring, pigmented lesions or sunburn which could interfere with the rating of efficacy parameters.
4. History of psoriasis unresponsive to topical treatments.
5. History of organ transplant requiring immunosuppression, HIV, or other immunocompromised state.
6. Use within 180 days prior to Baseline Visit of biologic treatment for psoriasis (e.g., infliximab, adalimumab, etanercept, ustekinumab, or alefacept).
7. Have received treatment for any type of cancer within 5 years of the Baseline Visit except for non-melanoma skin cancer and cervical cancer (in situ) are allowed within 1 year of the Baseline Visit.
8. Use within 60 days prior to the Baseline Visit of: 1) immunosuppressive drugs (e.g., tacrolimus, pimecrolimus), 2) systemic antipsoriatic treatment (e.g., methotrexate, cyclosporine, hydroxyurea) or 3) oral retinoids (e.g., acitretin, isotretinoin).
9. Use within 30 days prior to the Baseline Visit of: 1) systemic steroids, 2) PUVA therapy, 3) systemic anti-inflammatory agents (e.g., mycophenolate mofetil, sulfasalazine, 6-thioguanine), or 4) UVB therapy. Note: Inhaled, intraocular and intranasal steroids are allowed.
10. Use within 14 days prior to the Baseline Visit of: 1) topical antipsoriatic drugs (e.g., salicylic acid, anthralin, coal tar, calcipotriene), 2) topical retinoids (e.g., tazarotene, tretinoin) or 3) topical corticosteroids.
11. Subjects with known hypersensitivity to clocortolone pivalate or any component of Cloderm Cream.
12. Subjects who have participated in a study of an investigational drug 60 days prior to the Baseline Visit.
13. Subjects unable to comply with study requirements.
14. Female subjects who are pregnant (or planning to become pregnant) or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-10; Primary Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne M Fraser, PhD, Study Director — Promius Pharma
Locations (5):
- United States (5):
  - Radiant Research, Inc., Cincinnati, Ohio
  - Oregon Medical Research, Portland, Oregon
  - DermResearch, Inc., Austin, Texas
  - Research Across America, Dallas, Texas
  - Madison Skin and Research, Inc., Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Cloderm Cream: Cloderm (clocortolone pivalate) Cream 0.1%, twice daily for 28 days
  Cloderm Cream
Period: Overall Study
Arm/Group | Cloderm Cream
Started | 60
Completed | 57
Not Completed | 3
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cloderm Cream
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 55
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 60
Region of Enrollment [Number; unit: participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Investigator's Global Assessment (IGA)
Description: The proportion of subjects who demonstrate an IGA score of clear (0) or almost clear (1).
Time Frame: 28 days
Population: Intent to treat population, with LOCF for missing data
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Cloderm Cream
Number analyzed (Participants) | 60
percentage of subjects | 15 [8.1 to 26.1]

ADVERSE EVENTS:
Arm/Group | Cloderm Cream
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No report, abstract, oral presentation, or publication proposed by the Investigator/Institution in regard to Study shall be presented or published without the prior written consent of the Sponsor. Sponsor reserves the right to comment on and delay the proposed report, abstract, oral presentation, or publication and to revise as necessary to protect confidential information or intellectual property.